CLINICAL TRIAL: NCT02129608
Title: A Feasibility Pilot Comparing a Non-invasive Low Level Laser Therapy (LLLT) With Lorcaserin to Reduce Central Adiposity in Overweight Individuals.
Brief Title: Low Level Laser Treatment (LLLT) and Lorcaserin for Weight Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ivana Croghan, PhD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-002370
Record Dates: First submitted 2014-04-25; First posted 2014-05-02 (Estimated); Results first posted 2016-11-22 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-09

CONDITIONS: Overweight; Obese
Keywords: overweight; obese; central adiposity; Laser; lorcaserin; low level laser therapy; belviq
MeSH Terms: conditions — Overweight; Obesity; Obesity, Abdominal | interventions — Low-Level Light Therapy; lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LLLT (Active Comparator): Low Level Laser Therapy (LLLT) once a week for 12 weeks
  Interventions: Device: LLLT
- Lorcaserin (Active Comparator): locarserin monotherapy - 10 mg, twice daily for 12 weeks
  Interventions: Drug: Lorcaserin
- LLLT and Lorcaserin (Active Comparator): LLLT once a week for 12 weeks and 10 mg of Lorcaserin twice daily for 12 weeks
  Interventions: Device: LLLT; Drug: Lorcaserin

INTERVENTIONS:
Device: LLLT — The LLLT uses 6 diode laser heads - each emitting 17 mW output. Subject will receive 30 minutes of therapy in the frontal central area and 30 minutes of therapy in the back central area, once a week for 12 weeks.
  Other Names: Low Level Laser; Erchonia® Zerona™ 2.0 Laser
  Arms: LLLT; LLLT and Lorcaserin
Drug: Lorcaserin — 10 mg pills twice daily for 12 weeks.
  Other Names: Belviq
  Arms: LLLT and Lorcaserin; Lorcaserin

SUMMARY:
Currently in the United States about 97 million adults are considered obese, accounting for about 33% of the American adult population (compared to 22.9% in 1988). Obesity, defined as a body mass index of 30.0 or higher, is accountable for 44% of the diabetes, 23% of the ischemic heart disease and between 7% and 41% of certain cancers. The Erchonia® Zerona™ 2.0 Laser (which will be used in this study) has been approved by the FDA (K123237) as a non-invasive dermatological aesthetic treatment which can be used by individuals intending to reduce circumference of hips, waist, and thighs. Lorcaserin is a selective serotonin 2C (5-HT(2C)) receptor agonist. The exact mechanism of action is not known, but lorcaserin is believed to promote satiety and decrease food intake by activating 5-HT(2C) receptors on anorexigenic pro-opiomelanocortin neurons in the hypothalamus. Lorcaserin was approved by the FDA on June 2012 for weight management in people with a BMI of > 27 kg/m2 (overweight) when accompanied by a weigh-related condition such as type 2 diabetes or high blood pressure or in people with a BMI > 30 kg/m2 (obese). The purpose of this pilot study is to obtain preliminary data on: 1) effectiveness of the combination of LLLT and lorcaserin for reducing abdominal subcutaneous fat in overweight/obese individuals; 2) impact of LLLT on inflammatory biomarkers, blood sugar, and cholesterol.

DETAILED DESCRIPTION:
This study is being done to find out how effective Low Level Laser Therapy (LLLT - Erchonia® Zerona™ 2.0 Laser) is compared to Lorcaserin (Belviq®) in helping overweight people reduce their weight gain - especially in the central body region. Subjects will undergo 2 screening visits in which the investigators will take their medical and weight concern histories; and if found eligible, they will be randomized to one of three groups: 1) 12 weeks of LLLT, 2) 12 weeks of Lorcaserin, and 3) 12 weeks of a combination of both Lorcaserin and LLLT. Full study participation will last approximately 6 months and consists of 10 visits- 9 clinical and 1 phone call. During this study subjects will be provided with weight prevention counseling and be asked to complete 3 additional fasting blood draws. There will be one urine pregnancy test (for females only) at the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* be 18-70 years of age;
* have a body weight of greater than 50 kg (110 pounds);
* have a BMI 27-39.9 kg/m2;
* be weight concerned;
* be motivated to reduce their central adiposity;
* be able to participate fully in all aspects of the study;
* have understood and signed study informed consent.

Exclusion Criteria:

* have used weight loss medications or participated in a weight loss program within the past 30 days;
* are currently taking supplements known to affect weight, such as garcinia cambrogia.
* have had weight fluctuations of 20 pounds or more in the past 6 months (self-report);
* have an implanted device (including pacemaker or lap band) in the targeted area of LLLT;
* have an active untreated clinically significant psychiatric condition (psychosis, bipolar disorder, or depression);
* have used an investigational drug within 30 days of study enrollment;
* have a recent history (past 30 days) of alcohol or drug abuse or dependence;
* are currently pregnant or lactating, or are of child-bearing potential or are likely to become pregnant during the medication phase and are unwilling to use a reliable form of contraception;
* have a history of any major cardiovascular events including heart valve disease, cardiac arrhythmias, congestive heart failure, acute coronary syndrome, stroke, transient ischemic attack, or peripheral vascular disease;
* have current uncontrolled hypertension (systolic > 165 mm Hg or diastolic > 95 mm Hg) documented on 2 separate occasions;
* have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, lymphatic, respiratory, or metabolic disease (such as diabetes) or active cancer or are within 1 year of cancer remission;
* Prior surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery, etc.;
* medical, physical, or other contraindications for body sculpting/weight loss;
* current use of medication(s) known to affect weight levels/cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent;
* concurrently taking a serotonergic drug (selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MAOIs), triptans, bupropion, dextromethorphan, St. John's Wort). These drugs can be used to treat depression and/or migraines but are contraindicated with lorcaserin;
* any medical condition known to affect weight levels and/or to cause bloating or swelling;
* diagnosis of, and/or taking medication for, irritable bowel syndrome;
* active infection, wound or other external trauma to the areas to be treated with the laser;
* known photosensitivity disorder;
* are allergic to lorcaserin;
* current active cancer or currently receiving treatment for cancer; or
* have a known history of any condition or factor judged by the investigator to preclude participation in the study or which might hinder adherence;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T. Croghan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Croghan IT, Ebbert JO, Schroeder DR, Hurt RT, Hagstrom V, Clark MM. A randomized, open-label pilot of the combination of low-level laser therapy and lorcaserin for weight loss. BMC Obes. 2016 Sep 29;3:42. doi: 10.1186/s40608-016-0122-4. eCollection 2016. PMID 27708788
- See also: Related Info — http://bmcobes.biomedcentral.com/articles/10.1186/s40608-016-0122-4

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LLLT | Lorcaserin | LLLT and Lorcaserin
Started | 15 | 14 | 15
End of Treatment | 15 | 13 | 12
Completed | 15 | 13 | 12
Not Completed | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LLLT | Lorcaserin | LLLT and Lorcaserin | Total
Number analyzed (Participants) | 15 | 14 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 14 | 15 | 44
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (9.9) | 40.6 (11.5) | 45.4 (13.3) | 43.9 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 13 | 37
  Male | 2 | 3 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 14 | 14 | 15 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 15 | 14 | 15 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 15 | 44
Weight (in kgs) [Mean (Standard Deviation); unit: kg] | 96.0 (15.3) | 94.4 (16.2) | 90.3 (14.0) | 93.5 (15.0)
waist circumference (in cm) [Mean (Standard Deviation); unit: cm] | 105.3 (11.6) | 108.0 (15.7) | 100.9 (10.0) | 104.7 (12.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Waist Circumference
Description: The change in waist circumference from baseline to 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | LLLT | Lorcaserin | LLLT and Lorcaserin
Number analyzed (Participants) | 15 | 14 | 15
cm | -2.3 (4.1) | -6.0 (7.3) | -4.0 (5.5)
Statistical Analysis 1: Comparison: LLLT vs LLLT and Lorcaserin; Test type: Superiority or Other; p = 0.398, t-test, 2 sided
Statistical Analysis 2: Comparison: Lorcaserin vs LLLT and Lorcaserin; Test type: Superiority or Other; p = 0.436, t-test, 2 sided

2. Primary Outcome: Change in Weight
Description: The change in weight from baseline to 3 months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | LLLT | Lorcaserin | LLLT and Lorcaserin
Number analyzed (Participants) | 15 | 14 | 15
kg | -1.0 (4.4) | -3.7 (3.3) | -3.5 (3.6)
Statistical Analysis 1: Comparison: LLLT vs LLLT and Lorcaserin; Test type: Superiority or Other; p = 0.070, t-test, 2 sided
Statistical Analysis 2: Comparison: Lorcaserin vs LLLT and Lorcaserin; Test type: Superiority or Other; p = 0.950, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | LLLT | Lorcaserin | LLLT and Lorcaserin
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 2/14 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LLLT (N=15) | Lorcaserin (N=14) | LLLT and Lorcaserin (N=15)
dizziness (General disorders) | 0 (0) | 1 (1) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Low Blood Pressure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Tingling (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No